CLINICAL TRIAL: NCT04955288
Title: Research on Key Technologies and System Optimization of Early Warning and Resuscitation of Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-0420
Record Dates: First submitted 2021-06-20; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Emergencies
Keywords: 5G; Aortic Balloon Occlusion Catheter; Esophageal cooling device; Cardiopulmonary resuscitation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aortic balloon Assisted resuscitation group (Experimental): The aortic balloon-assisted resuscitation group uses aortic balloon occlusion technology on the basis of the traditional resuscitation mode, that is, when the cardiopulmonary resuscitation begins, the aortic balloon catheter is quickly punctured and inserted to the distal end of the aortic area I via ultrasound. (Septum level), then continue to inflate the balloon to block the aortic blood flow until the end of the cardiopulmonary resuscitation to deflate the balloon and remove the balloon catheter.
  Interventions: Procedure: Aortic balloon assisted resuscitation
- Traditional cardiopulmonary resuscitation group (Active Comparator): The traditional cardiopulmonary resuscitation group uses the traditional manual chest compression mode, that is, referring to the latest version of the cardiopulmonary resuscitation guidelines, manual chest compressions are performed under the monitoring of the compression quality feedback device to ensure that the compression depth is 5-6cm, the frequency is 100-120 times/min, Conditions such as a fixed compression position and sufficient chest wall rebound.
  Interventions: Procedure: Traditional cardiopulmonary resuscitation
- Esophageal cooling group (Experimental): The esophageal cooling group adopts a new transesophageal cooling method, that is, an esophageal cooling catheter is placed after resuscitation in patients with cardiac arrest, and then a small temperature-controlled water circulation system is continuously perfused with 4℃ cold water. After the patient's body temperature reaches the target temperature of 33℃, the temperature is adjusted Control the water circulation system to maintain the target body temperature of (33±0.5)°C for 24 hours, and then reheat to (37±0.5)°C normal body temperature at a rate of 0.25-0.5°C/h and maintain it for 24 hours.
  Interventions: Procedure: Esophageal cooling
- Traditional cooling group (Active Comparator): The traditional cooling group uses the traditional body surface ice blanket cooling method, that is, the patients with cardiac arrest lie on the temperature control blanket after resuscitation, and then use the ice blanket host to continuously infuse the temperature control blanket with 4℃ cold water, and wait until the patient's body temperature reaches the target temperature of 33℃ After that, adjust the ice blanket host to control the circulating water temperature to maintain the target body temperature of (33±0.5)°C for 24 hours, and then reheat to the normal body temperature of (37±0.5)°C at a rate of 0.25-0.5°C/h and maintain it for 24 hours.
  Interventions: Procedure: traditional cooling

INTERVENTIONS:
Procedure: Aortic balloon assisted resuscitation — On the basis of the traditional resuscitation mode, the aortic balloon occlusion technology is used, that is, at the same time when the cardiopulmonary resuscitation starts, the aortic balloon catheter is quickly punctured to the distal end of the aortic zone I (septum level) through ultrasound assistance, and then Continue to inflate the balloon to block the aortic blood flow until the end of the cardiopulmonary resuscitation to deflate the balloon and remove the balloon catheter.
  Arms: Aortic balloon Assisted resuscitation group
Procedure: Traditional cardiopulmonary resuscitation — Use the traditional manual chest compression mode, that is, refer to the latest version of the CPR Guidelines.
  Artificial chest compressions are performed under the monitoring of the pressure quality feedback device to ensure that the compression depth is 5-6cm, the frequency is 100-120 times/min, the compression position is fixed, and the chest wall fully rebounds.
  Arms: Traditional cardiopulmonary resuscitation group
Procedure: Esophageal cooling — The new transesophageal cooling method is adopted, that is, the esophageal cooling catheter is indwelled after resuscitation in patients with cardiac arrest, and then connected to a small temperature-controlled water circulation system to continuously infuse 4℃ cold water. After the patient's body temperature reaches the target temperature of 33℃, the temperature-controlled water circulation system is adjusted Maintain the target body temperature of (33±0.5)°C for 24 hours, and then rewarm to (37±0.5)°C normal body temperature at a rate of 0.25-0.5°C/h and maintain it for 24 hours.
  Arms: Esophageal cooling group
Procedure: traditional cooling — The traditional body surface ice blanket cooling method is adopted, that is, the patient with cardiac arrest lies on the temperature control blanket after resuscitation, and then uses the ice blanket host to continuously infuse the temperature control blanket with 4℃ cold water, and wait until the patient's body temperature reaches the target temperature of 33℃. The temperature of the circulating water is controlled by adjusting the ice blanket host to maintain the target body temperature of (33±0.5)°C for 24 hours, and then reheat to the normal body temperature of (37±0.5)°C at a rate of 0.25-0.5°C/h and maintain it for 24 hours.
  Arms: Traditional cooling group

SUMMARY:
Studies have shown that early prevention and warning of cardiac arrest, rapid implementation of high-quality cardiopulmonary resuscitation, and strengthening of organ function protection after resuscitation are the keys to reducing the occurrence of cardiac arrest and improving the prognosis of patients. However, there are still many problems in the field of cardiopulmonary resuscitation in my country: 1) lack of effective prevention and early self-rescue system for cardiac arrest; 2) traditional resuscitation techniques implemented in pre-hospital and emergency rooms and poor results; 3) organs after resuscitation Insufficient protection means and effects. In our early stage, focusing on the above key issues, the study found that 5G technology can help high-risk emergency events including early warning, early detection and first aid of cardiac arrest. Aortic balloon occlusion can significantly improve the effectiveness of cardiopulmonary resuscitation. Transesophageal and CRRT cooling Can significantly optimize the organ protection intensity of therapeutic hypothermia. On the basis of the preliminary work, this project will carry out the research and development and clinical application of a series of new technologies for cardiac arrest warning and resuscitation, and work hard to help with cardiac arrest. Early warning and treatment of cases provide a set of optimized diagnosis and treatment technical solutions, which has important scientific, clinical and social significance.

DETAILED DESCRIPTION:
1. During the period from January 2022 to December 2023, based on the early warning and emergency response system of cardiac arrest, real-time monitoring of the vital information of the recruited high-risk populations of cardiac arrest, and timely reporting of the above-mentioned populations with unstable vital signs Distribute early warning information, contact community doctors to provide medical assistance, 120 emergency centers for referrals, and hospitals to prepare for admission, etc., in order to reduce the occurrence of cardiac arrest in high-risk groups; ②January 2022-December 2023 During the period, when a cardiac arrest event occurred in the recruited population based on the above-mentioned system, the nearby social volunteers, community doctors, and 120 emergency centers were quickly activated. Rescue team members quickly went to rescue, and at the same time realized experts' real-time observation and guidance of on-site treatment scenes through the remote consultation system, and prepared for continuous treatment in the hospital, in order to improve the effect of resuscitation and treatment of cardiac arrest in high-risk populations; ③analyze the above Within 2 years of application of the system, the incidence of cardiac arrest and the outcome of early resuscitation and treatment in the recruited high-risk population.
2. Selected patients with cardiac arrest in our hospital from January 2022 to December 2023. Selection criteria: a. 18-75 years old, no gender limit; b. Advanced life support; c. Meet ethical requirements and sign informed consent. Exclusion criteria: a. Refusal of cardiopulmonary resuscitation; b. Indications of non-resuscitation for traumatic cardiac arrest; c. Patients with terminal malignant tumors or other diseases. The patients undergoing cardiac arrest were randomly divided into the traditional cardiopulmonary resuscitation group and the aortic balloon-assisted resuscitation group. The former adopts the traditional chest compression mode, and the latter uses aortic balloon blockade on the basis of the traditional resuscitation mode. Technology, compare the resuscitation effects of patients with cardiac arrest in our hospital within 2 years, such as the duration of cardiopulmonary resuscitation, the amount of adrenaline, the number of defibrillation, the success rate of resuscitation, the survival rate of admission, etc., to clarify that aortic balloon occlusion can improve the effectiveness of cardiopulmonary resuscitation Significant role in.
3. Selected patients with cardiac arrest in our hospital from January 2022 to December 2023. Selection criteria: a. 18 to 75 years old, no gender limit; b. return to spontaneous circulation; c. coma; d. meet ethical requirements and sign informed consent. Exclusion criteria: a. Cardiac arrest time> 10 min; b. Cardiopulmonary resuscitation time> 60 min; c. Hemodynamics need to be maintained by high-dose vasoactive drugs (adrenaline or norepinephrine dosage> 1μg/kg.min); d. The state of dying; e. Patients with advanced malignant tumors or other end-stage diseases. Cardiac arrest patients who had obtained spontaneous circulation were randomly divided into traditional cooling group and esophageal cooling group, respectively, as soon as possible after resuscitation, using body surface cooling blanket device and esophageal cooling device to implement sub-hypothermia, and compare the effect of low-temperature implementation in patients within 2 years, such as the start time, Target length, maintenance of low temperature, rewarming and other indicators, as well as clinical prognostic indicators such as multiple organ dysfunction, adverse events, ICU length of stay, total length of stay, immediate discharge and neurological prognosis and survival at 1, 3, and 6 months In order to clarify the strong protective effect of optimal implementation of therapeutic mild hypothermia through the esophagus on multiple organ damage after resuscitation.

ELIGIBILITY:
Inclusion Criteria:

18-75 years old Provide advanced life support Meet ethical requirements and sign informed consent return to spontaneous circulation coma

Exclusion Criteria:

Refusal of cardiopulmonary resuscitation Indications of non-resuscitation in the presence of traumatic cardiac arrest Patients with terminal malignant tumors or other diseases Cardiac arrest time>10min Cardiopulmonary resuscitation time>60min Hemodynamics need to be maintained by large doses of vasoactive drugs (adrenaline or norepinephrine dosage>1μg/kg.min) On the verge of Death status Patients with advanced malignant tumors or other end-stage diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
return of spontaneous circulation (ROSC) | 1-3 hours
  ROSC can be identified with the following three conditions: 1. arterial pulse can be reached; 2. effective ECG rhythm; 3. systolic blood pressure > 60 mmHg (1 mm Hg = 0.133 kPa).

OTHER OUTCOMES:
survival to discharge | 2 days
  whether patients survive to hospital discharge
survival to discharge without severe neurological impairment | 2 days
  defined as a CPC score of 1~2, which denotes survival with no more than moderate neurological disability with the ability to walk without assistance.
1-month survival without severe neurological impairment | 1 months
  patients who have survived for 1 month after cardiac arrest with a CPC score of 1~2
6-month survival without severe neurological impairment | 6 months
  patients who have survived for 6 months after cardiac arrest with a CPC score of 1~2
insertion-related complications | 2 days
  Whether esophageal mucosal injury,aortic injury,or some other complications occur in patients

CONTACTS AND LOCATIONS:
Overall Officials: Mao Zhang, PHD, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine & Institute of Emergency Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Hawkes C, Booth S, Ji C, Brace-McDonnell SJ, Whittington A, Mapstone J, Cooke MW, Deakin CD, Gale CP, Fothergill R, Nolan JP, Rees N, Soar J, Siriwardena AN, Brown TP, Perkins GD; OHCAO collaborators. Epidemiology and outcomes from out-of-hospital cardiac arrests in England. Resuscitation. 2017 Jan;110:133-140. doi: 10.1016/j.resuscitation.2016.10.030. Epub 2016 Nov 17. PMID 27865775
- [Background] Shao F, Li CS, Liang LR, Li D, Ma SK. Outcome of out-of-hospital cardiac arrests in Beijing, China. Resuscitation. 2014 Nov;85(11):1411-7. doi: 10.1016/j.resuscitation.2014.08.008. Epub 2014 Aug 20. PMID 25151546
- [Background] Weisfeldt ML, Becker LB. Resuscitation after cardiac arrest: a 3-phase time-sensitive model. JAMA. 2002 Dec 18;288(23):3035-8. doi: 10.1001/jama.288.23.3035. No abstract available. PMID 12479769
- [Background] Guidelines 2000 for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Part 6: advanced cardiovascular life support: section 1: Introduction to ACLS 2000: overview of recommended changes in ACLS from the guidelines 2000 conference. The American Heart Association in collaboration with the International Liaison Committee on Resuscitation. Circulation. 2000 Aug 22;102(8 Suppl):I86-9. doi: 10.1161/01.cir.102.suppl_1.i-86. No abstract available. PMID 10966665
- [Background] Laver S, Farrow C, Turner D, Nolan J. Mode of death after admission to an intensive care unit following cardiac arrest. Intensive Care Med. 2004 Nov;30(11):2126-8. doi: 10.1007/s00134-004-2425-z. Epub 2004 Sep 9. PMID 15365608
- [Background] Singh B, Zhang S, Ching CK, Huang D, Liu YB, Rodriguez DA, Hussin A, Kim YH, Chasnoits AR, Cerkvenik J, Muckala KA, Cheng A. Improving the utilization of implantable cardioverter defibrillators for sudden cardiac arrest prevention (Improve SCA) in developing countries: Clinical characteristics and reasons for implantation refusal. Pacing Clin Electrophysiol. 2018 Dec;41(12):1619-1626. doi: 10.1111/pace.13526. Epub 2018 Oct 31. PMID 30320410
- [Background] Xu F, Zhang Y, Chen Y. Cardiopulmonary Resuscitation Training in China: Current Situation and Future Development. JAMA Cardiol. 2017 May 1;2(5):469-470. doi: 10.1001/jamacardio.2017.0035. No abstract available. PMID 28297007
- [Background] Ringh M, Rosenqvist M, Hollenberg J, Jonsson M, Fredman D, Nordberg P, Jarnbert-Pettersson H, Hasselqvist-Ax I, Riva G, Svensson L. Mobile-phone dispatch of laypersons for CPR in out-of-hospital cardiac arrest. N Engl J Med. 2015 Jun 11;372(24):2316-25. doi: 10.1056/NEJMoa1406038. PMID 26061836
- [Background] Kleinman ME, Brennan EE, Goldberger ZD, Swor RA, Terry M, Bobrow BJ, Gazmuri RJ, Travers AH, Rea T. Part 5: Adult Basic Life Support and Cardiopulmonary Resuscitation Quality: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S414-35. doi: 10.1161/CIR.0000000000000259. No abstract available. PMID 26472993
- [Background] Brooks SC, Anderson ML, Bruder E, Daya MR, Gaffney A, Otto CW, Singer AJ, Thiagarajan RR, Travers AH. Part 6: Alternative Techniques and Ancillary Devices for Cardiopulmonary Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S436-43. doi: 10.1161/CIR.0000000000000260. No abstract available. PMID 26472994
- [Background] Aufderheide TP, Pirrallo RG, Yannopoulos D, Klein JP, von Briesen C, Sparks CW, Deja KA, Kitscha DJ, Provo TA, Lurie KG. Incomplete chest wall decompression: a clinical evaluation of CPR performance by trained laypersons and an assessment of alternative manual chest compression-decompression techniques. Resuscitation. 2006 Dec;71(3):341-51. doi: 10.1016/j.resuscitation.2006.03.021. Epub 2006 Oct 27. PMID 17070644
- [Background] Zhu N, Chen Q, Jiang Z, Liao F, Kou B, Tang H, Zhou M. A meta-analysis of the resuscitative effects of mechanical and manual chest compression in out-of-hospital cardiac arrest patients. Crit Care. 2019 Mar 27;23(1):100. doi: 10.1186/s13054-019-2389-6. PMID 30917840
- [Background] Tang W, Weil MH, Noc M, Sun S, Gazmuri RJ, Bisera J. Augmented efficacy of external CPR by intermittent occlusion of the ascending aorta. Circulation. 1993 Oct;88(4 Pt 1):1916-21. doi: 10.1161/01.cir.88.4.1916. PMID 8403337
- [Background] Gedeborg R, Silander HC, Rubertsson S, Wiklund L. Cerebral ischaemia in experimental cardiopulmonary resuscitation--comparison of epinephrine and aortic occlusion. Resuscitation. 2001 Sep;50(3):319-29. doi: 10.1016/s0300-9572(01)00350-1. PMID 11719162
- [Background] Tsurukiri J, Akamine I, Sato T, Sakurai M, Okumura E, Moriya M, Yamanaka H, Ohta S. Resuscitative endovascular balloon occlusion of the aorta for uncontrolled haemorrahgic shock as an adjunct to haemostatic procedures in the acute care setting. Scand J Trauma Resusc Emerg Med. 2016 Feb 9;24:13. doi: 10.1186/s13049-016-0205-8. PMID 26861070
- [Background] Chaudery M, Clark J, Morrison JJ, Wilson MH, Bew D, Darzi A. Can contrast-enhanced ultrasonography improve Zone III REBOA placement for prehospital care? J Trauma Acute Care Surg. 2016 Jan;80(1):89-94. doi: 10.1097/TA.0000000000000863. PMID 26683394
- [Background] Daley J, Morrison JJ, Sather J, Hile L. The role of resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct to ACLS in non-traumatic cardiac arrest. Am J Emerg Med. 2017 May;35(5):731-736. doi: 10.1016/j.ajem.2017.01.010. Epub 2017 Jan 12. PMID 28117180
- [Background] Brede JR, Lafrenz T, Klepstad P, Skjaerseth EA, Nordseth T, Sovik E, Kruger AJ. Feasibility of Pre-Hospital Resuscitative Endovascular Balloon Occlusion of the Aorta in Non-Traumatic Out-of-Hospital Cardiac Arrest. J Am Heart Assoc. 2019 Nov 19;8(22):e014394. doi: 10.1161/JAHA.119.014394. Epub 2019 Nov 11. PMID 31707942
- [Background] Xu J, Shen P, Gao Y, Xia S, Liu S, Li Z, Zhou G, Xu Y, Zhang M. The Effects of the Duration of Aortic Balloon Occlusion on Outcomes of Traumatic Cardiac Arrest in a Porcine Model. Shock. 2019 Sep;52(3):e12-e21. doi: 10.1097/SHK.0000000000001235. PMID 30052583
- [Background] Neumar RW, Nolan JP, Adrie C, Aibiki M, Berg RA, Bottiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT Jr, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Vanden Hoek T. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A consensus statement from the International Liaison Committee on Resuscitation (American Heart Association, Australian and New Zealand Council on Resuscitation, European Resuscitation Council, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Asia, and the Resuscitation Council of Southern Africa); the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; and the Stroke Council. Circulation. 2008 Dec 2;118(23):2452-83. doi: 10.1161/CIRCULATIONAHA.108.190652. Epub 2008 Oct 23. No abstract available. PMID 18948368
- [Background] Nolan JP, Soar J, Cariou A, Cronberg T, Moulaert VR, Deakin CD, Bottiger BW, Friberg H, Sunde K, Sandroni C. European Resuscitation Council and European Society of Intensive Care Medicine Guidelines for Post-resuscitation Care 2015: Section 5 of the European Resuscitation Council Guidelines for Resuscitation 2015. Resuscitation. 2015 Oct;95:202-22. doi: 10.1016/j.resuscitation.2015.07.018. No abstract available. PMID 26477702
- [Background] Lascarrou JB, Merdji H, Le Gouge A, Colin G, Grillet G, Girardie P, Coupez E, Dequin PF, Cariou A, Boulain T, Brule N, Frat JP, Asfar P, Pichon N, Landais M, Plantefeve G, Quenot JP, Chakarian JC, Sirodot M, Legriel S, Letheulle J, Thevenin D, Desachy A, Delahaye A, Botoc V, Vimeux S, Martino F, Giraudeau B, Reignier J; CRICS-TRIGGERSEP Group. Targeted Temperature Management for Cardiac Arrest with Nonshockable Rhythm. N Engl J Med. 2019 Dec 12;381(24):2327-2337. doi: 10.1056/NEJMoa1906661. Epub 2019 Oct 2. PMID 31577396
- [Background] Schock RB, Janata A, Peacock WF, Deal NS, Kalra S, Sterz F. Time to Cooling Is Associated with Resuscitation Outcomes. Ther Hypothermia Temp Manag. 2016 Dec;6(4):208-217. doi: 10.1089/ther.2016.0026. Epub 2016 Oct 19. PMID 27906641
- [Background] Chenoune M, Lidouren F, Adam C, Pons S, Darbera L, Bruneval P, Ghaleh B, Zini R, Dubois-Rande JL, Carli P, Vivien B, Ricard JD, Berdeaux A, Tissier R. Ultrafast and whole-body cooling with total liquid ventilation induces favorable neurological and cardiac outcomes after cardiac arrest in rabbits. Circulation. 2011 Aug 23;124(8):901-11, 1-7. doi: 10.1161/CIRCULATIONAHA.111.039388. Epub 2011 Aug 1. PMID 21810660
- [Background] Deye N, Cariou A, Girardie P, Pichon N, Megarbane B, Midez P, Tonnelier JM, Boulain T, Outin H, Delahaye A, Cravoisy A, Mercat A, Blanc P, Santre C, Quintard H, Brivet F, Charpentier J, Garrigue D, Francois B, Quenot JP, Vincent F, Gueugniaud PY, Mira JP, Carli P, Vicaut E, Baud FJ; Clinical and Economical Impact of Endovascular Cooling in the Management of Cardiac Arrest (ICEREA) Study Group. Endovascular Versus External Targeted Temperature Management for Patients With Out-of-Hospital Cardiac Arrest: A Randomized, Controlled Study. Circulation. 2015 Jul 21;132(3):182-93. doi: 10.1161/CIRCULATIONAHA.114.012805. Epub 2015 Jun 19. PMID 26092673
- [Background] Polderman KH, Noc M, Beishuizen A, Biermann H, Girbes AR, Tully GW, Seidman D, Albertsson PA, Holmberg M, Sterz F, Holzer M. Ultrarapid Induction of Hypothermia Using Continuous Automated Peritoneal Lavage With Ice-Cold Fluids: Final Results of the Cooling for Cardiac Arrest or Acute ST-Elevation Myocardial Infarction Trial. Crit Care Med. 2015 Oct;43(10):2191-201. doi: 10.1097/CCM.0000000000001158. PMID 26196354
- [Background] Xu J, Jin X, Chen Q, Wu C, Li Z, Zhou G, Xu Y, Qian A, Li Y, Zhang M. Faster Hypothermia Induced by Esophageal Cooling Improves Early Markers of Cardiac and Neurological Injury After Cardiac Arrest in Swine. J Am Heart Assoc. 2018 Nov 6;7(21):e010283. doi: 10.1161/JAHA.118.010283. PMID 30608213
- [Background] Xu J, Chen Q, Jin X, Wu C, Li Z, Zhou G, Xu Y, Qian A, Li Y, Zhang M. Early Initiation of Continuous Renal Replacement Therapy Induces Fast Hypothermia and Improves Post-Cardiac Arrest Syndrome in a Porcine Model. Shock. 2019 Oct;52(4):456-467. doi: 10.1097/SHK.0000000000001276. PMID 30335673